CLINICAL TRIAL: NCT01155609
Title: L-lysine in the Treatment of Oral Mucositis in Head and Neck Cancer Patients- A Pilot Study
Brief Title: L-lysine in Treating Oral Mucositis in Patients Undergoing Radiation Therapy With or Without Chemotherapy For Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 7101; NCI-2010-01425 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-06-29; First posted 2010-07-02 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Mucositis; Oral Complications of Chemotherapy; Oral Complications of Radiation Therapy; Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Basal Cell Carcinoma of the Lip; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage I Adenoid Cystic Carcinoma of the Oral Cavity; Stage I Basal Cell Carcinoma of the Lip; Stage I Lymphoepithelioma of the Nasopharynx; Stage I Lymphoepithelioma of the Oropharynx; Stage I Mucoepidermoid Carcinoma of the Oral Cavity; Stage I Salivary Gland Cancer; Stage I Squamous Cell Carcinoma of the Hypopharynx; Stage I Squamous Cell Carcinoma of the Larynx; Stage I Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage I Squamous Cell Carcinoma of the Nasopharynx; Stage I Squamous Cell Carcinoma of the Oropharynx; Stage I Verrucous Carcinoma of the Larynx; Stage I Verrucous Carcinoma of the Oral Cavity; Stage II Adenoid Cystic Carcinoma of the Oral Cavity; Stage II Basal Cell Carcinoma of the Lip; Stage II Lymphoepithelioma of the Nasopharynx; Stage II Lymphoepithelioma of the Oropharynx; Stage II Mucoepidermoid Carcinoma of the Oral Cavity; Stage II Salivary Gland Cancer; Stage II Squamous Cell Carcinoma of the Hypopharynx; Stage II Squamous Cell Carcinoma of the Larynx; Stage II Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage II Squamous Cell Carcinoma of the Nasopharynx; Stage II Squamous Cell Carcinoma of the Oropharynx; Stage II Verrucous Carcinoma of the Larynx; Stage II Verrucous Carcinoma of the Oral Cavity; Stage III Adenoid Cystic Carcinoma of the Oral Cavity; Stage III Basal Cell Carcinoma of the Lip; Stage III Lymphoepithelioma of the Nasopharynx; Stage III Lymphoepithelioma of the Oropharynx; Stage III Mucoepidermoid Carcinoma of the Oral Cavity; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Adenoid Cystic Carcinoma of the Oral Cavity; Stage IV Basal Cell Carcinoma of the Lip; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Lymphoepithelioma of the Oropharynx; Stage IV Mucoepidermoid Carcinoma of the Oral Cavity; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity
MeSH Terms: conditions — Mucositis; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Lysine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supportive care (oral complications management) (Experimental): Patients receive L-Lysine PO QD until completion of radiotherapy and resolution of mucositis in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: quality-of-life assessment; Procedure: management of therapy complications; Dietary Supplement: L-lysine

INTERVENTIONS:
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Procedure: management of therapy complications — Discontinue supplement; treat symptomatically
  Other Names: complications of therapy, management of
Dietary Supplement: L-lysine — Given PO
  Other Names: L-lysine monohydrate; lysine monohydrate

SUMMARY:
This pilot clinical trial studies L-lysine in treating oral mucositis in patients undergoing radiation therapy with or without chemotherapy for head and neck cancer. L-lysine may lessen the severity of oral mucositis, or mouth sores in patients receiving radiation therapy with or without chemotherapy for head and neck cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete response rate, decrease in severity, and time to complete response of oral mucositis related to head and neck cancer irradiation and chemotherapy after using L-lysine supplementation daily.

SECONDARY OBJECTIVES:

I. To determine the functional impact of use of L-lysine for oral mucositis on daily life as measured by the Functional Life Index-Cancer (FLIC) Questionnaire total score.

OUTLINE:

Patients receive L-lysine orally (PO) once daily (QD) until completion of radiotherapy and resolution of mucositis in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up weekly until mucositis resolves.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or pathologically proven cancer of the oropharynx, lip, oral cavity, larynx, hypopharynx, nasopharynx, and salivary glands
* Predicted life expectancy greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Renal function with a calculated creatinine clearance of 55 ml/min or greater, per Cockcroft-Gault formula
* Patients undergoing radiation therapy with or without concurrent chemotherapy
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria

* Use of illicit drugs, alcohol abuse, or tobacco abuse during treatment
* Subjects may not be receiving other investigational agents
* Inability or unwillingness to comply with radiation therapy and chemotherapy regimens
* Inability or unwillingness to take daily L-Lysine supplementation as prescribed
* Use of arginine supplementation
* History of renal failure or compromise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Decrease in mucositis severity and time to complete response | Weekly post-treatment until Grade 0 mucositis is achieved
  Complete Response will be documented by complete resolution of oral mucositis, as defined by the Radiation Therapy Oncology Group (RTOG) grading scale. If the true percent of patients that respond is 20%, we will have a 90% chance of seeing at least 1 patient in 10 with a response. If none of the 10 patients show significant improvement in time to response, then we can be 90% confident that the true rate of significant improvement is less than 20%.

SECONDARY OUTCOMES:
Improvement in quality of life | Weekly post-treatment until Grade 0 mucositis is achieved

CONTACTS AND LOCATIONS:
Overall Officials: Upendra Parvathaneni, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States